CLINICAL TRIAL: NCT00389077
Title: A Phase IIA Trial of Two Schedules of Perifosine
Brief Title: Trial of Two Schedules of Perifosine for Patients With Solid Tumors or Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Perifosine 207
Record Dates: First submitted 2006-10-16; First posted 2006-10-18 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2011-11

CONDITIONS: Tumors; Lymphomas
Keywords: perifosine; solid tumors; lymphomas; anticancer agent
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — perifosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Perifosine Daily Dose (Experimental): Daily dose perifosine 50 mg.
  Interventions: Drug: Perifosine
- Perifosine Twice Daily Dose (Experimental): Twice daily dose perifosine 50 mg.
  Interventions: Drug: Perifosine

INTERVENTIONS:
Drug: Perifosine — Perifosine 50 mg tablets
  Other Names: D-21266; KRX-0401

SUMMARY:
This is a study of the drug perifosine for patients who have no standard treatment options. This study is designed to identify which cancer types respond to perifosine, and determine which regimen of perifosine is most effective in each one. Patients with either solid tumors or with lymphomas for whom this protocol represents reasonable or optimal treatment will be randomized to receive either perifosine 100 mg daily or 900 mg weekly until disease progression. Based on currently available data it is anticipated that these doses should be easily tolerated by most patients.

DETAILED DESCRIPTION:
This is an exploratory phase IIA trial with unique elements of design and patient selection with an aim to:

* Identify responsive tumor types that were not predicted from preclinical and Phase I studies,
* Determine if tumors are more likely to stabilize than shrink, and
* Identify a dose with almost no toxicity.
* To determine whether response (or stabilization) can be observed on either a daily or weekly schedule, or both. Since the efficacy goal of the study is to look for any evidence of activity with perifosine, the daily and weekly arms will be combined when assessing response.
* Response to therapy will be based on either tumor regression (objective response, partial or complete) OR stabilization of disease.

It is not anticipated that this study will provide "proof of principle" regarding the use of perifosine or serve as a pivotal trial for regulatory purposes. Information obtained from this study will be used to design additional trials that will be more definitive in nature.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically or cytologically confirmed diagnosis of either a lymphoma or solid tumor for which there is no established therapy that, in the opinion of the treating physician, will prolong the patient's survival or have a larger net effect on the patient's quality of life.
* The physician must believe that the patient's course and the growth rate of the tumor are such that the patient would feel comfortable continuing treatment for at least 12 weeks even if there were a transient period of modest tumor growth (defined as less than 30%) during the first weeks following the initiation of perifosine treatment.
* Patients must have a life expectancy of more than 6 months.
* Patients must not be eligible for any other available perifosine study.
* In general, patients should have received no more than two prior cytotoxic chemotherapy regimens for metastatic disease.
* Patients may have measurable or non-measurable disease. If the outcome for a patient is to be based on response using Response Evaluation Criteria in Solid Tumors (RECIST) criteria, the patient must have at least one measurable lesion that can be accurately measured in at least one dimension and fit one of the following criteria: longest diameter >= 20 mm using conventional techniques or >= 10 mm with spiral computed tomography (CT) scan. The dimensions of all target lesions that will be used to determine objective response along with the date of last measurement and the method of measurement (e.g. physical examination, spiral CT, conventional CT) must be recorded on the enrollment form prior to the patient's first treatment.
* If the outcome for a patient is to be based on an increase in time to progression, the following will apply:

  * The time to progression on the systemic treatment administered just prior to enrollment in this trial must be carefully documented and should be 12 weeks or more.
  * There must have been a baseline tumor evaluation in which all sites of likely metastases, based on signs and symptoms, were evaluated at the beginning of this pre-protocol baseline time interval. (A total body CT scan or magnetic resonance imaging [MRI] will usually suffice but are not required to meet this criterion).
  * During the 12+ weeks in which the patient was progression-free, there must have been no symptoms or signs of new metastases that warranted an evaluation, undertaken or not.
  * Progression of prior metastases or the appearance of new metastases must be documented at the end of the progression-free 12+ week period.
  * This prior progression-free interval must be recorded on the enrollment case report form prior to the patient's first treatment.
* Patients should have a performance status of 0 to 1 according to the ECOG criteria.
* Patients must have adequate organ and marrow function. Adequate organ and marrow function are described below.

  * hematocrit (HCT) >= 28% (with or without growth factor support)
  * creatinine <= 2.5 mg/dl
  * total bilirubin <= 1.5x upper limit of normal
  * transaminase <= 2.5x upper limit of normal
* Patients must have recovered from acute toxicity related to prior therapy including surgery or radiotherapy, excluding alopecia.
* Patients with breast cancer or prostate cancer who discontinue endocrine therapy prior to entry into this study must wait for a minimum of 1 month and then be reassessed for a withdrawal response prior to starting perifosine. However, it is not a requirement that endocrine therapies be discontinued.
* Patients must be able to ingest oral medications or to obtain them through a gastrostomy tube.
* Patients must be at least 18 years of age
* Patients must have ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Rapidly progressing disease, as defined by progression within 12 weeks of initiation of the previous regimen
* Patients receiving any other investigational agents or devices
* Patients who have recently (within 8 weeks) begun a new cancer treatment (e.g., bisphosphonates) that will be continued concomitantly with perifosine
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to perifosine (miltefosine or edelfosine)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection and psychiatric illness/social situations that would limit compliance with study requirements
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with perifosine.
* Patients with a history of unstable or newly diagnosed angina pectoris, recent myocardial infarction (within 6 months of enrollment), or New York Heart Association class II-IV congestive heart failure
* Female patients who are pregnant or lactating are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2005-01; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (PR + CR) | Evaluated every 12 weeks
  To determine for each disease category the proportion of patients treated with perifosine who experience a favorable outcome, defined as a complete or partial response; a 50% increase in progression-free survival compared to patient's latest treatment regimen for metastatic disease, or stabilization of disease.

SECONDARY OUTCOMES:
To Show that doses will be each sufficiently and tolerated | From date of randomization
  To show that daily 50 mg daily and 50 mg twice-daily doses are each sufficiently well tolerated to ensure good compliance in future studies of these two regimens
To obtain plasma levels | Every treatment cycle
  To obtain perifosine plasma levels in a subset of patients to evaluate variability in drug uptake between patients, and to correlate plasma levels with outcomes to insure good compliance in future studies of these two regimens

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Goggins, MD, Study Chair — Fox Valley Hematology and Oncology SC, Appleton

REFERENCES:
- [Result] 1) Journal of Clinical Oncology, 2009 ASCO Annual Meeting Proceedings (Post-Meeting Edition). Vol 27, No 15S (May 20 Supplement), 2009: e15505 / For HCC ( hepatic / sub-population) 2) Journal of Clinical Oncology, 2007 ASCO Annual Meeting Proceedings (Post-Meeting Edition). Vol 25, No 18S (June 20 Supplement), 2007: 15622 / For RCC (renal / sub-population)